CLINICAL TRIAL: NCT05989971
Title: The Effect of Continuous Renal Replacement Therapy on the Efficiency of Extracorporeal CO2 Removal
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, deputy director, Southeast University, China
Other Study IDs: 20230731
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Failure With Hypercapnia
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extracorporeal carbon dioxide removal combined with continuous renal replacement therapy: extracorporeal carbon dioxide removal combined with continuous veno-venous hemofiltration or continuous veno-venous hemodialysis.CVVH and CVVHD set-up: predilution 30 ml/kg/h, dialysate dose 30 ml/kg/h, ultrafiltration rate was equal to the total rate of substitution fluid infusion.
  Interventions: Other: continuous renal replacement therapy

INTERVENTIONS:
Other: continuous renal replacement therapy — continuous veno-venous hemofiltration or continuous veno-venous hemodialysis set-up: predilution 30 ml/kg/h, dialysate dose 30 ml/kg/h, ultrafiltration rate was equal to the total rate of substitution fluid infusion

SUMMARY:
In the design of extracorporeal carbon dioxide removal (ECCO2R) combined with continuous renal replacement therapy (CRRT) equipment, in model of continuous veno-venous hemofiltration (CVVH) , the HCO3- concentration in the pre membrane lung blood is diluted by the replacement solution, and a decrease in HCO3- leads to a decrease in PCO2. On the other hand, in continuous veno-venous hemodialysis (CVVHD), HCO3- in post membrane blood will exchange interaction. The exchange results of HCO3- determine the impact of CVVHD on the CO2 removal efficiency of the ECCO2R combined CRRT system. This study aims to investigate the effects of CVVH and CVVHD on in vitro CO2 clearance efficiency.

DETAILED DESCRIPTION:
In the design of extracorporeal carbon dioxide removal (ECCO2R) combined with continuous renal replacement therapy (CRRT) equipment, the pre dilution replacement solution for continuous veno-venous hemofiltration (CVVH) enters the extracorporeal bloodstream upstream of the membrane lung, so the HCO3- concentration in the pre membrane lung blood is diluted by the replacement solution. HCO3- and dissolved CO2 are in a dynamic and rapid equilibrium state, and a decrease in HCO3- leads to a decrease in PCO2. On the other hand, in continuous veno-venous hemodialysis (CVVHD), the blood after the membrane needs to undergo material exchange with the dialysate through a filter. The dialysate is usually HCO3- with normal plasma concentration, so HCO3- in post membrane blood will exchange interaction. The exchange results of HCO3- determine the impact of CVVHD on the CO2 removal efficiency of the ECCO2R combined CRRT system. This study aims to investigate the effects of CVVH and CVVHD on in vitro CO2 clearance efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Using Extracorporeal carbon dioxide removal combined with continuous renal replacement therapy
* 18 years ≤ age ≤ 85 years;

Exclusion Criteria:

* Severe hemodynamic instability (increased dosage of vasoactive drugs or MAP ≤ 65mmHg within two hours);
* Severe electrolyte deficiency (including severe hyponatremia (blood sodium<130mmol/L) and hypokalemia (blood potassium<3.0mmol/L));
* Participate in other intervention studies within 30 days;
* Do not consent this research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: using Extracorporeal carbon dioxide removal combined with continuous renal replacement therapy
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
extracorporeal CO2 removal rate | after 30min of continuous renal replacement therapy
  extracorporeal CO2 removal rate was calculated as the difference of total CO2 content before membrane lung and after hemofilter, and normalized to an inlet PCO2 of 45 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, Study Director — Zhongda Hospital
Locations (1):
- Ling Liu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No